CLINICAL TRIAL: NCT01599728
Title: Urocortins 2 & 3-Effects on Forearm Arterial Blood Flow in Patients With Heart Failure
Brief Title: Effect of Urocortins in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: UcnHFP2
Record Dates: First submitted 2012-05-14; First posted 2012-05-16 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Heart Failure; Endothelium
Keywords: Urocortin 2; Urocortin 3; Forearm venous occlusion plethysmography; Heart failure; Endothelium; Substance P
MeSH Terms: conditions — Heart Failure | interventions — Urocortins; Substance P

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with heart failure (Other): Assessing the response to infusion of intra-arterial Urocortin 2, 3 and Substance P in patients with heart failure
  Interventions: Drug: Urocortin 2, Urocortin 3 and Substance P
- Healthy controls (Other): Assessing response to intra-arterial infusions of Urocortin 2, 3 and Substance P in age and sex-matched healthy volunteers as controls.
  Interventions: Drug: Urocortin 2, Urocortin 3 and Substance P

INTERVENTIONS:
Drug: Urocortin 2, Urocortin 3 and Substance P — After a 20-min infusion of intra-arterial saline, ascending doses of Urocortin 2 (3.6, 12 and 36 pmol/min [15, 50 and 150 ng/min] to achieve estimated end-organ concentrations of 0.6, 2 and 6 µg/L, respectively), Urocortin 3 1200, 3600 and 12000 pmol/min (5, 15 and 50 micrograms/min) [to achieve estimated end-organ concentrations of 199, 600 and 2000 micrograms/L respectively] and substance P (a control endothelium-dependent vasodilator that evokes endogenous t-PA release [2, 4 and 8 pmol/min]) will be administered intra-arterially.
  Baseline blood samples will be taken at the start of the study for full blood count, cholesterol, glucose, renal function Bilateral venous blood samples will be taken at baseline, immediately before the start of Ucn2/Ucn3 infusion and at the end of each dose of Ucn2/Ucn3 for subsequent measurement of plasma Ucn 2 and 3 concentrations and other hormones.

SUMMARY:
Despite modern advances in treatment, heart failure continues to carry a poor prognosis with high morbidity and mortality rates. Hence, there remains a major interest in the development of novel therapeutic agents for this debilitating condition. Urocortins have recently shot into limelight with their potential role in the pathophysiology and treatment of heart failure.

Recent studies by the investigators group (REC no: 09/S1103/41) have confirmed that Urocortin 2 and 3 are potent arterial vasodilators, the effects of which are reproducible and well tolerated in healthy male volunteers. Previous studies using heart failure models in animals1-7, as well studies in heart failure patients (Urocortin 2), suggest that there is great scope for Urocortins as novel biomarkers and as potential therapeutic agents in heart failure. With this in mind, the investigators wish to study the local vasomotor effects of these peptides in greater detail in patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

Patients with heart failure:

1. Patients with stable heart failure (NYHA class II-IV) on maximum tolerated doses of an ACE inhibitor and beta-blocker for at least 3 months.
2. Baseline echocardiographic parameters (echo performed within last 12 months) at recruitment: ejection fraction (EF) <35%, left ventricular end dimension >5.5cm and fractional shortening <20%
3. Age 18-80 years (inclusive) at recruitment

Healthy volunteers:

* Age and sex-matched healthy volunteers

Exclusion Criteria:

1. Lack of informed consent
2. Age <18 years and > 80 years
3. Current involvement in a clinical trial
4. Systolic blood pressure >190 mmHg or <90 mmHg, untreated malignant arrhythmias
5. Haemodynamically significant valvular heart disease
6. Severe or significant co-morbidity including bleeding diathesis, renal or hepatic failure
7. History of anaemia
8. Recent infective/inflammatory condition
9. Recent blood donation (prior 3 months)
10. Women of child bearing potential

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow | 3 hours
  Difference between forearm blood flow in response to doses of Ucn2, Ucn3 and Substance P between heart failure patients and healthy controls.

SECONDARY OUTCOMES:
Absolute forearm blood flow | 3 hours
  Absolute forearm arterial blood flow in response to Ucn2, Ucn3 and Substance P.

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD, FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Wellcome Trust Clinical Research Facility, Royal Infirmary of Edinburgh, Edinburgh, United Kingdom